CLINICAL TRIAL: NCT07016048
Title: Facial Scanning and Computerized Tomography as Aids in Single-tooth Rehabilitation Planning
Brief Title: Digital Technologies in Dental Rehabilitation Planning.
Acronym: PHDSL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1409
Record Dates: First submitted 2025-05-20; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Digital Technologies in Dental Rehabilitation Planning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Static occlusion (Placebo Comparator): Use IOS + DPhotos - Set up the models and do a diagnostic waxing done only with static occlusion, without a virtual articulator (as the laboratories commonly do).
  Interventions: Procedure: Try-in of one crown test with a digital wax-up (per group)
- Virtual articulator (standard values) (Active Comparator): Use IOS + DPhotos - Set up the models do a diagnostic waxing in the virtual articulator arbitrarily (without CBCT and FS) - with the program's default and standard values.
  Interventions: Procedure: Try-in of one crown test with a digital wax-up (per group)
- Virtual articulator with CBCT and FS (standard values) (Active Comparator): Use IOS + DPhotos + CBCT + FS - Set up the models and do a diagnostic waxing in the virtual articulator (with CBCT and FS) - with the program's default and standard values.
  Interventions: Procedure: Try-in of one crown test with a digital wax-up (per group)
- Programmed virtual articulator (Active Comparator): Use IOS + DPhotos + CBCT + FS - Set up the models and do a diagnostic waxing in the virtual articulator (with CBCT and FS) - with the articulator programmed for the patient - through dynamic scans.
  Interventions: Procedure: Try-in of one crown test with a digital wax-up (per group)

INTERVENTIONS:
Procedure: Try-in of one crown test with a digital wax-up (per group) — In a CAD/CAM software, we will integrate IOS, CBCT, and FS data into the virtual environment, and it will be possible the articulation of virtual models.
  The digital wax-up for the preparation of the crown will be designed by the prosthodontist and then adjusted based on the occlusion obtained in each of the groups.
  The steps of clinical procedure are:
  1. - In the first appointment, the patients mention their smile concerns, and the dentist evaluate and diagnoses.
  2. - Digital impressions, and a model of the teeth will be done.
  3. - Diagnostic wax-up, where dentist and dental laboratory plan the wax-up on the study models.
  4. - Diagnostic mock-up, where dentist transfers the diagnostic wax-up to the patient's mouth.
  We will evaluate the volumetric difference between the diagnostic wax-ups obtained in each group.
  After each mock-up, a questionnaire will be delivered to the patients in order to assess patients's aesthetics and comfort self-perception, using a numeric scale.

SUMMARY:
The goal of this clinical trial is to evaluate the influence of Facial Scan (FS) and cone beam computed tomography (CBCT) in the prosthodontic treatment planning in patients who require rehabilitation with a single crown.

After collecting the patients, at the first appointment, data collection will be carried out, including: an intraoral scan (digital impressions), intraoral and extraoral photographs, CBCT, and facial scanning.

At the following appointment, a mock-up will be performed. The purpose of the mock-up is to preview the expected smile outcome before beginning the oral rehabilitation treatment.

After each mock-up, patients will be asked to complete a questionnaire designed to evaluate their self-perception of comfort and aesthetics.

Additionally, after each mock-up, the clinician will assess occlusal contacts (the bite) and record the time required for adjustments to achieve a comfortable occlusion for the patient.

The main questions it aims to answer are:

* How does the patient perceive comfort and aesthetics during the rehabilitation process?
* What is the influence of using a virtual articulator on diagnostic waxing accuracy?
* How does integrating facial scanning (FS) and cone-beam computed tomography (CBCT) affect current digital workflows involving a virtual articulator?
* What impact does the programming of the virtual articulator have on treatment planning outcomes?

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the influence of Facial Scan (FS) and cone beam computed tomography (CBCT) in the prosthodontic treatment planning in patients who require rehabilitation with a single crown, with aims:

i) assessing patient's comfort and aesthetics self-perception; ii) evaluate the influence of a virtual articulator in a diagnostic waxing; iii) evaluate the influence of implementation of FS and CBCT to the current digital procedure with a virtual articulator; iv) evaluate the influence of programming the virtual articulator.

Data collection will be carried out in participants, including: an intraoral scan (digital impressions), intraoral and extraoral photographs (DPhotos), CBCT, and facial scan.

In a CAD/CAM software, we will integrate IOS, CBCT, and FS data into the virtual environment, and it will be possible the articulation of virtual models.

The digital wax-up for the preparation of the crown will be designed by the prosthodontist and then adjusted based on the occlusion obtained in each of the groups.

The design and occlusal adjustment of the crown will carry out in four different ways, separating them into the following groups:

* Group 1: IOS + DPhotos - Diagnostic waxing done only with static occlusion, without a virtual articulator (as the laboratories commonly do).
* Group 2: IOS + DPhotos - Set up the models in the virtual articulator arbitrarily (without CBCT and FS) - with the program's default and standard values.
* Group 3: IOS + DPhotos + CBCT + FS - Set up the models in the virtual articulator (with CBCT and FS) - with the program's default and standard values.
* Group 4: IOS + DPhotos + CBCT + FS - Set up the models in the virtual articulator (with CBCT and FS) - with the articulator programmed for the patient - through dynamic scans.

For the representation of the Group 4, we will program a virtual articulator by modifying the values of the condylar guidance angles, in order to realize the changes that could occur just by modifying them. During the study, we plan to program the articulator with dynamic scans of each patient. These dynamic scans will result in individually customised condylar guidance angles.

Four crown tests will be produced, one for each group, to enable them to be tried out on participants (like a mock-up).

Participants enrolled in this study will be randomly allocated in the 4 groups, with a computer-generated randomization list (https://www.randomizer.org/).

Allocation concealment will be performed using sealed and opaque numbered envelopes which were opened by the dentist immediately before the mock-up.

All the procedures will be performed by one experienced clinician.

The steps of clinical procedure are:

Step 1 - In the first appointment, the patients mention their smile concerns, and the dentist evaluate and diagnoses.

Step 2 - Digital impressions, and a model of the teeth will be done. Step 3 - Diagnostic wax-up, where dentist and dental laboratory plan the wax-up on the study models.

Step 4 - Diagnostic mock-up, where dentist transfers the diagnostic wax-up to the patient's mouth.

We will evaluate the volumetric difference (in micrometers) before and after occlusal adjustments, in each group; and the volumetric difference between the diagnostic wax-ups obtained in each group.

After each mock-up, a questionnaire will be delivered to the patients in order to assess patients's aesthetics and comfort self-perception, using a numeric scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require rehabilitation with a single crown;
* The tooth to be rehabilitated must have an opponent to test the occlusion.

Exclusion Criteria:

* The tooth to be rehabilitated must does not have an opponent to test the occlusion;
* Edentulous patient;
* Incapable of understanding and/or giving consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Differences before and after occlusal adjustments | From enrollment to the end of treatment (8 weeks)
  The primary outcome is the volumetric difference (in micrometers) before and after occlusal adjustments, in each group.

SECONDARY OUTCOMES:
Patients's aesthetics and comfort self-perception | From enrollment to the end of treatment (8 weeks)
  The secondary outcome measure is the patient's comfort and aesthetics self-perception - with questionnaires, using a numerical scale.

OTHER OUTCOMES:
Occlusion differences between diagnostic wax-ups | From enrollment to the end of treatment (8 weeks)
  Other outcome is the volumetric difference (in micrometers) between the diagnostic wax-ups obtained in each group.

IPD SHARING:
Plan to Share IPD: Yes